CLINICAL TRIAL: NCT05195788
Title: Investigating the Impact of Cardiac Rehabilitation on Brain Activity and Cognition in Adults With Congenital Heart Disease
Brief Title: Cardiac Rehabilitation in Congenital Heart Disease: Effects on Brain and Cognitive Functions
Acronym: CongeNIRS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Montreal Heart Institute (Other)
Responsible Party: Principal Investigator, Louis Bherer, Associate Scientific Director, Direction of Prevention, Montreal Heart Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MHI 2022-3019
Record Dates: First submitted 2021-12-13; First posted 2022-01-19 (Actual); Last update posted 2023-11-21 (Actual); Status verified 2023-11

CONDITIONS: Congenital Heart Disease; Congenital Heart Defects
Keywords: Congenital Heart Disease; Congenital Heart Defects; Brain; fNIRS; Cognition; Cardiac rehabilitation; Exercise
MeSH Terms: conditions — Heart Defects, Congenital; Motor Activity | interventions — Cardiac Rehabilitation

STUDY DESIGN:
Intervention Model Description: The CongeNIRS study uses the prospective, randomised, open-label, blinded end-point (PROBE) design.
  The participation in this study is expected to be three months and two weeks, comprising three months of physical training and 2 weeks of testing (baseline and three months, one week each).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Participants assigned to the Intervention group will undergo a cardiac rehabilitation program. The program will combine individualized aerobic and muscle strengthening exercises, comprising three sessions per week to be conducted in person at the EPIC center and at home, for a duration of three months. All sessions will be prepared by a certified kinesiologist.
  Interventions: Behavioral: Cardiac rehabilitation
- Control (No Intervention): Participants assigned to the control group will be encouraged to remain at the usual level of physical activity for the duration of the study. At the end of the study, they will gain free access to the same cardiac rehabilitation program provided to the intervention group.

INTERVENTIONS:
Behavioral: Cardiac rehabilitation — The cardiac rehabilitation program is based on 3/week exercise training's sessions including aerobic and muscle building exercises. All exercises are individualized, supervised by a certified kinesiologist at the research center, and in line with the latest recommendations for physical activity in individuals with congenital heart disease. Participants are encouraged to do a minimum of 1 supervised session per week at the research center and may, with the agreement of the cardiologist and the kinesiologist, do the other training sessions at home (hybrid program). The characteristics of the activities are recorded with a heart rate sensor. Each session lasts a maximum of 60 minutes in total and includes approximately 30 minutes of aerobic exercise, and approximately 20 minutes of muscle strengthening exercises, with 5 to 10 minutes of warm-up and cool-down.
  Arms: Intervention

SUMMARY:
The proposed trial is designed to evaluate the effect of an individualised cardiac rehabilitation program, consisting of aerobic and muscle strengthening exercises, on brain activity and cognitive functions in adults with congenital heart disease

DETAILED DESCRIPTION:
Thanks to advances in medical research, individuals born with heart defects (Congenital Heart Disease: CHD), are now 95% more likely to reach adulthood, with around 250,000 adults with CHD currently living in Canada. CHD-related diseases and conditions are extremely common in the adult CHD population, and undermine the successes achieved by medical research. For example, compared to healthy peers, adults with CHD are between 3 to 6 times more likely to experience heart accidents or develop other heart conditions during lifetime. Adults with CHD also have more health problems, and have between 1.5 and 2 increased risk of precocious cognitive decline and dementia. Better lifestyle choices and management of medical risk factors play a crucial role in preventing such problems and in increasing the quality of life of those living with CHD. In this regard, physical activity has been suggested as one of the most cost-effective methods for decreasing mortality and incidence of cardiovascular diseases related to CHD. An increasing body of studies have shown that both physical activity and exercise training improve physical and mental health in adults with CHD, who typically tend to be less active than healthy adults. Although physical activity and exercise training have been shown to enhance cognition and brain activity in individuals with other cardiovascular diseases, such effects in CHD are yet to be investigated.

In the present project, the impact of a cardiac rehabilitation program on brain activity and on cognitive functions will be explored in adults with moderate and severe forms of CHD. The 3-month intervention will include an individualised program consisting of combined aerobic and muscle strengthening exercises provided by certified kinesiologists, to be completed at the research center and at home (hybrid program). Brain imaging technology (fNIRS) will be used to measure changes in brain activity related to the intervention. The benefits on cognitive functions, such as attention, executive functions and memory, will be measured with standardized neuropsychological tests before and after the intervention. The results of this project will contribute to a better understanding of the many benefits of exercise training in individuals with CHD, and will lay the foundations for optimal interventions, targeted to prevent CHD-related conditions and impairments.

ELIGIBILITY:
Inclusion Criteria:

* being able to read, understand and sign the information and consent form;
* being aged 18 or more at the time of consent;
* having a diagnosis of congenital heart disease with moderate or severe risk;
* being referred to the EPIC center in cardiovascular rehabilitation;
* being able to perform a maximal cardiopulmonary stress test and an exercise training program in accordance with current recommendations for cardiovascular rehabilitation;
* having Internet access.

Exclusion Criteria:

* recent major cardiovascular events or interventions <3 months;
* uncontrolled mental or psychiatric disorder in the last 6 months;
* genetic syndromes affecting cognition;
* excessive alcohol consumption (> 15 drinks / week);
* current participation in other clinical trials;
* contraindication to stress testing and / or physical training;
* severe intolerance to physical exercise.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2022-02-07 (Actual); Primary Completion 2024-04 (Estimated); Study Completion 2024-04 (Estimated)

PRIMARY OUTCOMES:
Change in brain hemodynamics | Baseline, post-intervention at 3 months
  Neurovascular coupling (Stroop task). This component will be investigated at the cortical level using functional near infrared spectroscopy (fNIRS), and measured in changes in hemodynamics (oxygenated hemoglobin concentration).

SECONDARY OUTCOMES:
Changes in general cognitive functioning | Baseline, post-intervention at 3 months
  Cognitive performance. This component will be investigated using the Montreal Cognitive Assessment test.
Changes in episodic memory | Baseline, post-intervention at 3 months
  Memory performance. This component will be investigated using the Rey Auditory Verbal Learning test.
Changes in executive functions | Baseline, post-intervention at 3 months
  Cognitive performance. This component will be investigated using tests of executive functions (n-back, Trail Making Test, dual task, Stroop), measured in accuracy (composite Z-score).
Changes in processing speed | Baseline, post-intervention at 3 months
  Cognitive performance. This component will be investigated using tests of executive functions (Trail Making Test, dual task, Stroop), measured in reaction time (composite Z-score).

OTHER OUTCOMES:
Changes in cardiorespiratory fitness | Baseline, post-intervention at 3 months
  Maximal incremental cardiopulmonary exercise test (VO2 max).
Changes in cardiac hemodynamic | Baseline, post-intervention at 3 months
  Cardiac output will be measured continuously at rest and during exercise (L/min).

CONTACTS AND LOCATIONS:
Overall Officials: Louis Bherer, PhD, Principal Investigator — EPIC Center of the Montreal Heart Institute
Locations (1):
- EPIC Center of the Montreal Heart Institute, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Tran D, Maiorana A, Ayer J, Lubans DR, Davis GM, Celermajer DS, d'Udekem Y, Cordina R. Recommendations for exercise in adolescents and adults with congenital heart disease. Prog Cardiovasc Dis. 2020 May-Jun;63(3):350-366. doi: 10.1016/j.pcad.2020.03.002. Epub 2020 Mar 19. PMID 32201288
- [Background] Li X, Chen N, Zhou X, Yang Y, Chen S, Song Y, Sun K, Du Q. Exercise Training in Adults With Congenital Heart Disease: A SYSTEMATIC REVIEW AND META-ANALYSIS. J Cardiopulm Rehabil Prev. 2019 Sep;39(5):299-307. doi: 10.1097/HCR.0000000000000420. PMID 31343584
- [Background] Tran DL, Maiorana A, Davis GM, Celermajer DS, d'Udekem Y, Cordina R. Exercise Testing and Training in Adults With Congenital Heart Disease: A Surgical Perspective. Ann Thorac Surg. 2021 Oct;112(4):1045-1054. doi: 10.1016/j.athoracsur.2020.08.118. Epub 2020 Dec 4. PMID 33285131